CLINICAL TRIAL: NCT06086873
Title: A Randomised Clinical Trial Investigating Effect of Implant Surface Characteristic on Crestal Marginal Bone Loss, Inflammatory Response and Aesthetic Outcomes: Novel Gradient Anodized and Sandblasted Large-grit Acid-etched Implant Surfaces
Brief Title: Investigating Implant Surface Effect on Osseointegration: NGA vs. ModSLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160995; IRAS:329055 (Registry Identifier: IRAS)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NGA Implant (Experimental): NGA Implant (NobelActive TiUltraNP, Nobel Biocare AG, Switzerland)
  Interventions: Device: Implant Type
- BLX implant (BLX) modSLA Surface (Experimental): BLX implant (BLX) modSLA Surface (BLX, SLActive, Roxolid, Institut Straumann AG, Switzerland)
  Interventions: Device: Implant Type
- TLX implant (TLX) modSLA Surface (Experimental): TLX implant (TLX) modSLA Surface (TLX, SLActive, Roxolid, Institut Straumann AG, Switzerland).
  Interventions: Device: Implant Type

INTERVENTIONS:
Device: Implant Type — Patients enrolled in the study will be allocated to one of three implant groups:
  * Group 1: NGA Implant (NobelActive TiUltraNP, Nobel Biocare AG, Switzerland)
  * Group 2: BLX implant (BLX) modSLA Surface (BLX, SLActive, Roxolid, Institut Straumann AG, Switzerland)
  * Group 3: TLX implant (TLX) modSLA Surface (TLX, SLActive, Roxolid, Institut Straumann AG, Switzerland).

SUMMARY:
This study aims to characterise the stability of crestal bone levels one year after loading, the associated aesthetic outcomes, immunological response, prosthodontic outcomes as well as overall patient reported outcome measures for modSLA (SLActive, Institut Straumann AG, Switzerland) and NGA (TiUltraNP, Nobel Biocare AG, Switzerland) dental implants.

DETAILED DESCRIPTION:
Ultra-hydrophilic SLActive (modSLA) implants have been extensively studied in pre-clinical and clinical studies, demonstrating their pro-osteogenic nature and long-term maintenance of facial bone and aesthetics.

A novel multi-zone novel gradient anodized (NGA) hydrophilic surface (TiUltra) has recently been introduced to clinical practice. Pre-clinical studies have demonstrated that the smoother coronal aspect achieved stable soft tissue adhesion.

In clinical practice, prosthetically driven implant placement, particularly in the anterior maxilla, may result in a buccal dehiscence that is commonly treated with guided bone regeneration (GBR). Currently no studies have been published investigating differences between these commercially available implant surfaces (modSLA, NGA).

This prospective, single centre randomised clinical trial will recruit 39 patients who require a single tooth extraction in the anterior maxilla for a Type IIc implant placement.

Patients enrolled in the study will be allocated to one of three implant groups:

* Group 1: NGA Implant (NobelActive TiUltraNP, Nobel Biocare AG, Switzerland)
* Group 2: BLX implant (BLX) modSLA Surface (BLX, SLActive, Roxolid, Institut Straumann AG, Switzerland)
* Group 3: TLX implant (TLX) modSLA Surface (TLX, SLActive, Roxolid, Institut Straumann AG, Switzerland).

This study aims to characterise the stability of crestal bone levels one year after loading, the associated aesthetic outcomes, immunological response, prosthodontic outcomes as well as overall patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 years old,
* Gender: male and female.
* Patient must be able and willing to follow study procedures and instructions and have capacity to provide informed consent.
* Patient must require tooth extraction of a maxillary first premolar or single-rooted anterior tooth as the result of caries, endodontic failure or trauma
* The extraction site must have adjacent teeth present.
* Adjacent teeth with no evidence of interdental bone loss

Exclusion Criteria:

* Systemic disease that can interfere with dental implant therapy (e.g. uncontrolled diabetes)
* 2 adjacent teeth requiring extraction
* Greater than one wall of the socket missing - assessed at time of extraction
* Any contraindications for oral surgical procedures
* Any known systemic disease affecting bone metabolism (e.g. Cushing's syndrome, Crohn's disease, rheumatoid arthritis, osteoporosis, diabetes type I and uncontrolled diabetes type II), systemic infections or recent surgical procedures within 30 days of study initiation;
* Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine, calcium antagonists and cyclosporine) or bone metabolism (e.g. bisphosphonates, hormone replacement therapy, immunosuppressants) within 1 month before baseline visit;
* HIV or viral hepatitis;
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene;
* History of local irradiation therapy in the head-neck region
* Mucosal diseases (e.g. erosive lichen planus)
* Current untreated periodontitis or gingivitis. In particular probing depths of >4mm on one of the teeth immediately adjacent to the extraction site
* Untreated acute endodontic lesions
* Current smokers (have smoked within 3 months of study onset)
* Any known systemic disease affecting bone metabolism (e.g. Cushing's syndrome, Crohn's disease, rheumatoid arthritis, osteoporosis, diabetes type I and uncontrolled diabetes type II), systemic infections or recent surgical procedures within 30 days of study initiation;
* Self-reported alcoholism or chronic drug abuse;
* Patients suffering from a known psychological disorder or with limited mental capacity or language skills such that study information could not be understood,
* Non-compliant patients, vulnerable individuals or those unable to understand written or verbal communication and give consent.
* Pregnant or breastfeeding patients
* Involvement in current research or recent involvement in any research prior to recruitment
* Full-mouth bleeding (BOP) and plaque (PI) scores >30% or sites with periodontal pocket depth >5 mm at the completion of the pre-treatment phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Coronal Facial Bone Maintenance | 1 Year post loading
  A numerical comparison of coronal facial bone thickness between the groups. CBCT scans will be compared to quantify the linear changes in crestal bone thickness at the coronal aspect of the implant (shoulder of NGA and BLX implants and rough-smooth transition of TLX implant).

SECONDARY OUTCOMES:
Aesthetic Outcome | 1 Year post loading
  - A numerical comparison of the three groups from an objective aesthetic scale derived from a panel of 2 dentists.
Patient Satisfaction | 1 Year post loading
  - A numerical comparison of the patient satisfaction between the three groups derived from an analysis of patient questionnaires (Likert Scales).
Patient Satisfaction- Aesthetics | 1 Year post loading
  - A numerical comparison of the aesthetic merit between the three groups derived from an analysis of patient questionnaires (Likert scales)
Primary Stability | 1 Year post loading
  A numerical comparison of primary stability measurement of the three groups (IT, RFA).
Immunological Response | Pre-surgery to 12 Weeks post surgery
  - A numerical and qualitative comparison of inflammatory profiles derived from peripheral blood of the three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Dental Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No